CLINICAL TRIAL: NCT06297655
Title: A Phase III Clinical Study Evaluating the Efficacy and Safety of On-demand Treatment and Perioperative Replacement Therapy With Recombinant Human Coagulation Factor VIII for Injection in Treated Severe Hemophilia A
Brief Title: A Clinical Study of Recombinant Human Coagulation Factor VIII for Injection in Patients With Severe Hemophilia A
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Nanjing Shunxin Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQG202-III-01
Record Dates: First submitted 2024-03-01; First posted 2024-03-07 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Recombinant human activated coagulation factor Ⅷ for injection (Experimental): Each subject in this study receive on-demand treatment with recombinant human coagulation factor VIII for injection for 180 days, with an increase in medication frequency based on the relief after medication.
  Interventions: Drug: Recombinant human activated coagulation factor VIII for injection

INTERVENTIONS:
Drug: Recombinant human activated coagulation factor VIII for injection — Recombinant human coagulation factor VIII for injection is a recombinant DNA product with functional characteristics comparable to endogenous factor VIII.

SUMMARY:
This study is a single arm, open, multicenter clinical trial in which the previous treated severe hemophilia A patients receive recombinant human coagulation factor VIII for injection to evaluate the efficacy and safety of on-demand treatment in the event of new bleeding events. If evaluable surgical cases occur, the overall efficacy and safety of recombinant human coagulation factor VIII for injection as a replacement therapy for severe hemophilia A PTPs during the perioperative period will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* The subjects voluntarily joined this study, signed an informed consent form, and had good compliance;
* Age: ≥ 12 years old and ≤ 65 years old (when signing the informed consent form, if it is a minor, parents should sign on behalf of it);
* Severe hemophilia A (coagulation factor VIII activity<1%), with exposure days (ED) of no less than 150 days prior to factor VIII (recombinant coagulation factor VIII or plasma derived coagulation factor VIII) treatment; Surgical patients need to have undergone at least 2 surgeries (including major surgeries) and plan to undergo elective surgery at the same time;
* The subjects must be HIV negative or have a viral load of < 200 particles/μ, HIV positive patients with l or < 400000 copies/ml.
* At baseline, no inhibitors were detected, and there was no history of Factor VIII inhibitor antibody formation (Bethesda method detection < 0.6 BU/ml, test result record required);
* Subjects of childbearing age who agree to take effective contraceptive measures throughout the entire trial period and continue until 28 days after the last medication.

Exclusion Criteria:

* Known congenital or acquired hemorrhagic diseases other than hemophilia A;
* The subjects have used or planned to receive immunosuppressive treatments such as prednisone, cyclophosphamide, and cyclosporine in the week prior to enrollment, and are allowed to use inhaled or topical corticosteroids;
* Those who are known or suspected to have hypersensitivity reactions to the investigational drug, including human embryonic kidney cell protein;
* Significant liver and kidney dysfunction, including alanine aminotransferase (ALT) and aspartate aminotransferase (AST) > 5 upper limit of normal (ULN), and serum creatinine >1.5 ULN;
* Hemoglobin < 60 g/L;
* Expected to receive other drugs for the treatment of hemophilia A within 72 hours before the first administration (such as recombinant factor VIII, blood derived factor VIII, desmopressin, cryoprecipitate, plasma, etc.), or those who have used long-acting hemophilia A drugs for less than 5 half-lives before the first administration;
* Used within 14 days before the first administration or planned to use anticoagulants or antiplatelet drugs for treatment during clinical trials;
* Within 6 months prior to the first administration, use of Emicizumab;
* Serious cardiovascular and cerebrovascular diseases occurring within 6 months prior to the first administration, including but not limited to cerebral hemorrhage, cerebral infarction, unstable angina, malignant arrhythmia, acute myocardial infarction, congestive heart failure (New York Heart Association cardiac function classification ≥ III), and hypertension (systolic blood pressure ≥ 160 mmHg or diastolic blood pressure 100 mmHg) that is poorly controlled despite treatment with one or more antihypertensive drugs;
* Participated in clinical trials of other drugs within 30 days prior to screening, or last used investigational drug with less than 5 half-lives;
* Alcohol abuse, drug abuse, mental disorders, and intellectual disabilities.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
The proportion of on-demand treatment improvement for newly occurring bleeding events | For each new bleeding event, assessed within 72 hours after initial treatment
  Evaluate the hemostatic efficacy of the patient after each new bleeding event (including new bleeding events during visits and new bleeding events during home treatment), and calculate the proportion of improvement as excellent+good to the total number of on-demand treatment evaluations.
Activity recovery | 15 minutes after infusion
  The activity of Recombinant human coagulation factor VIII measured at 15 minutes after infusion minus the baseline Recombinant human coagulation factor VIII activity divided by the expected improvement in Recombinant human coagulation factor VIII activity, which reflects the improvement in Recombinant human coagulation factor VIII levels after infusion.

SECONDARY OUTCOMES:
The proportion of effective surgical hemostasis | Within 72 hours after surgery
  Assess the hemostatic efficacy of injecting recombinant human coagulation factor VIII during and after surgery. The effective ratio is the proportion of excellent or good to the total times of the surgical evaluation of hemostatic efficacy
Annualized bleeding rate (ABR) | Up to 180 days.
  Including spontaneous and traumatic bleeding, as well as total bleeding; ABR can be calculated using the following formula: bleeding frequency/(treatment period days/365.25).
The incidence of Less Han Expected Thermal Effect | For each new bleeding event, assessed within 24 hours after initial treatment
  Without the influence of confounding factors, continuously infuse Recombinant human coagulation factor VIII twice within 24 hours for on-demand treatment, with no response to the same bleeding event.
The injection times of recombinant human coagulation factor VIII | Up to 180 days.
  The injection times of recombinant human coagulation factor VIII for each new bleeding event.
The dosage of recombinant human coagulation factor VIII | Up to 180 days.
  The dosage of recombinant human coagulation factor VIII (including average and total doses) for each new bleeding event
Changes of Haemophilia Joint Health Score before and after on-demand treatment | Up to 180 days.
  The scale assesses the functional status of the six major joints of the elbow, knee, and ankle, including: joint swelling, swelling duration, muscle atrophy, muscle strength, joint friction, joint pain, joint extension, joint flexion Degree decline, overall gait, etc.
Changes of Quality of Life Assessment before and after on-demand treatment | Up to 180 days.
  Quality of Life Assessment is a general questionnaire designed to measure health status on a scale of 0-100 with the higher value representing a better outcome and record the participants' current health state in 5 domains mobility, selfcare, usual activities, pain, anxiety.

CONTACTS AND LOCATIONS:
Locations (11):
- China (11):
  - Anhui Provincial Hospital, Hefei, Anhui
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Henan Tumor Hospital, Zhengzhou, Henan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Nanjing Drug Tower Hospital, Nanjing, Jiangsu
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - Hematology Hospital of Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality
  - The Second Affiliated Hospital of Kunming Medical University, Kunming, Yunnan